CLINICAL TRIAL: NCT05278325
Title: Improved Treatment Course for Patients With Migraine and Tension-type Headache
Acronym: TeII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Louise Carlsen, PhD, MD, Danish Headache Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H18008942
Record Dates: First submitted 2022-02-23; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Migraine; Tension-Type Headache
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone Intervention (Experimental): Two planned phone call by health care professionals after 8 and 16 weeks adjusting acute and preventive treatment
  Interventions: Other: Telephone intervention
- Business as usual (No Intervention): No planned phone calls

INTERVENTIONS:
Other: Telephone intervention — Two planned phone call between clinical controls
  Arms: Telephone Intervention

SUMMARY:
The purpose of the study is to improve treatment for newly referred patients with migraine and tension-type headache to the Danish Headache Center.

All patients will recieve an electronic questionnaire just before the first visit concerning their current and previous history of headache and headache treatment.

Half of them will enter a special telephone-intervention (TeII) program with two planned phone-calls after 8 and 16 weeks from first visit. The other half of patients will follow the normal follow-up program.

All patients will be seen by a headache specialist after 6 months and will be asked to fill in a follow-up electronic questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Migraine and/or tension-type headache

Exclusion Criteria:

* Other headache diagnoses, including cluster headache, medication overuse-headache, other secondary headaches, trigeminal neuralgia.
* Included in clinical trials at the DHC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Change in preventive headache medication | From baseline to six months
  Difference in number of patients with change in preventive headache medication in the two groups
Change in acute headache medication | From baseline to six months
  Difference in number of patients with change in acute headache medication in the two groups

SECONDARY OUTCOMES:
Change in headache frequency | From baseline to six months
  Difference in change of headache days per month between the two groups
Change in migraine frequency | From baseline to six months
  Difference in change of migraine days per month between the two groups
Change in Headache Under response to Treatment (HURT-8) score | From baseline to six months
  Difference in change in HURT-8 scale between the two groups
Change in Insomnia Severity Index (ISI) score | From baseline to six months
  Difference in change in ISI score between the two groups
Change in Hospitality Anxiety Depression Scale (HADS) score | From baseline to six months
  Difference in change in HADS between the two groups
Change in patient satisfaction score | At six months
  Difference in change in patient satisfaction score (five questions focusing on treatment course) between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Henrik W Schytz, Ass Prof, Study Chair — Rigshospitalet-Glostrup, Afdeling for Hjerne- og Nervesygdomme
Locations (1):
- Danish Headache Center, Glostrup Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No